CLINICAL TRIAL: NCT01229137
Title: Physiological Response to Exercise: Sensor Evaluation at Specified Exertions
Acronym: PRE-SENSE
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PRE-SENSE; G100110 (Other: FDA)
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Right Ventricular Cohort: Right Ventricle wtih SRD-1 conversion
  Interventions: Device: SRD-1 conversion
- Left Ventricular Cohort: Left Ventricle with SRD-1 conversion
  Interventions: Device: SRD-1 conversion
- Right Atrium Cohart: Right atrium cohort with SRD-1 conversion
  Interventions: Device: SRD-1 conversion

INTERVENTIONS:
Device: SRD-1 conversion

SUMMARY:
Assessment of sensor parameter in patients with heart failure.

DETAILED DESCRIPTION:
Evaluate the correlation of specific sensor parameters with clinical reference measurements in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* COGNIS CRT-D model N119 or N120, functional bipolar leads: RA, RV, and LV lead all implanted for a minimum of 30 days
* Prescribed to optimal pharmacologic therapy for heart failure for at least 30 days prior to enrollment
* Age 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Documented HF decompensation, as defined by a hospitalization or greater than a doubling of baseline diuretic dose due to worsening HF, within the last 3 months
* Patients who are pacemaker dependent
* Creatinine ≥ 2.5 mg/dL test within the last 3 months
* Requires assistance walking, for example a cane or walker
* Have an atrial tachyarrhythmia that is permanent or persistent
* Have moderate to severe chronic pulmonary disease as defined by FEV1 < 55% predicted
* Documented life expectancy of less than 6 months
* Patients at an unreasonable risk of not being able to reach the investigational center in case of an emergency, per physician discretion
* Enrolled in any concurrent study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with an implanted CRT-D
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Bank, M.D., Principal Investigator — United Heart and Vascular Center
Locations (14):
- United States (14):
  - Cardiovascular Associates of Northeast Arkansas, Jonesboro, Arkansas
  - Regional Cardiology Consultants, Sacremento, California
  - Danbury Hospital, Danbury, Connecticut
  - Heart and Vascular Institute of Florida, Clearwater, Florida
  - Genesis Medical Center, Davenport, Iowa
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - St. John's Hospital and Medical Center, Detroit, Michigan
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cardiovascular Research Institure, LLC, Canton, Ohio
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - Tyler Cardiovascular Associates, Tyler, Texas
  - Thomas Bunch, Murray, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia